CLINICAL TRIAL: NCT01497106
Title: Effects of Calorie Restriction on Accumulation of Old, Modified Proteins in Abdominally Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-006181
Record Dates: First submitted 2011-12-16; First posted 2011-12-22 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; Abdominal obesity; Calorie restriction
MeSH Terms: conditions — Insulin Resistance; Obesity, Abdominal | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie restriction (Experimental): Participants will work with the CRU dietetics staff to plan a diet that will result in their losing 1-2 pounds per week over 16 weeks.
  Interventions: Behavioral: Calorie Restriction
- Control (Active Comparator): Participants will continue their normal living for entire time of the study, totaling 16 weeks.
  Interventions: Behavioral: Control (normal living)

INTERVENTIONS:
Behavioral: Calorie Restriction — Participants will work with the CRU dietetics staff to plan a diet that will result in their losing 1-2 pounds per week over 16 weeks. They will wear an accelerometer to track there activity during these weeks.
  Arms: Calorie restriction
Behavioral: Control (normal living) — Participants will continue their normal living for entire time of the study. They will be asked to wear an accelerometer for the next 16 weeks and check in weekly at the CRU to exchange accelerometers.
  Arms: Control

SUMMARY:
This study is being done to understand the effects of calorie restriction and weight loss on muscle protein metabolism in adult men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI will be between 30 kg/m2 - 38 kg/m2 and waist circumference for women ≥ 88 cm and men ≥ 104 cm
* Age 45 to 65 years.
* Male and Female

Exclusion Criteria:

* Active coronary artery disease
* BMI < 30 kg/m2 Participation in structured exercise (>2 times per week for 30 minutes or longer)
* Smoking
* Medications known to affect muscle metabolism (beta blockers)
* Renal failure (serum creatinine > 1.5mg/dl)
* Chronic active liver disease (AST and ALT > 3 times normal)
* Fasting blood glucose > 126 mg/dl
* Anti-coagulant therapy (warfarin/heparin)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis from baseline to 16 weeks | Measured at week 0 (baseline) and week 16
  The investigators will determine the rate of incorporation of stable isotope amino acid tracers in skeletal muscle protein on average resting muscle protein synthesis rate (% new muscle protein per hour) and will be performed at baseline and 16 weeks after caloric restriction or control diet.

SECONDARY OUTCOMES:
Change in insulin sensitivity from 0 (baseline) and 16 weeks | Measured at week 0 (baseline) and week 16
  The investigators will determine insulin sensitivity at week 0 (baseline) and 16 weeks into caloric restriction or control diet. The measurement is made by hyperinsulimic euglycemic clamp and reported as μmol per kilogram of fat free mass of infused glucose needed to maintain glycemia.

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States